CLINICAL TRIAL: NCT05465161
Title: An Ex-Vivo Human Model Study for Proof of Concept, Usability, Reproducibility, Radio-Opacity and Marker Retention
Brief Title: STING MARK Universal Fiducial Marker System
Acronym: StingMark
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CE 21.203
Record Dates: First submitted 2022-02-28; First posted 2022-07-19 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- StingMark Fiducial Marker (Experimental): Device insertion will occur with the designated needles and through the appropriate organ-specific route and imaging guidance. Multiple STING-MARK fiducials will be inserted. Plain film x-rays in 3 planes of the organs with the marker inserted will be taken and recorded.
  Interventions: Device: Sting Mark Fiducial Marker

INTERVENTIONS:
Device: Sting Mark Fiducial Marker — Device insertion will occur with the designated needles and through the appropriate organ-specific route and imaging guidance. Multiple STING-MARK fiducials will be inserted. Plain film x-rays in 3 planes of the organs with the marker inserted will be taken and recorded.

SUMMARY:
Currently available fiducial marker and fiducial insertion strategies are rudimentary, imprecise, not compatible with multiple insertion catheters/needles and are overall unreliable. STING-MARK device is the first universal, fully detachable and non-premounted radiopaque fiducial device system. Allowing biopsy prior to insertion, STING-MARK is easily and reliably delivered through-the-needle to the tumor, in order to accurately pinpoint its location for image-guided therapies. This study aims at establishing proof of concept for STING-MARK, by demonstrating its usability, reproducibility, radio-opacity and retention in a variety of clinically-relevant ex vivo organ samples.

DETAILED DESCRIPTION:
Patients undergoing surgical resection of solid organs at the CHUM or recipients of solid organ transplantation will be approached for consent into the study protocol. Human solid organs that are being removed for either elective surgery or transplantation will be removed in the standard manner and sent to the pathology laboratory as in the typical situation following removal. After the pathology team finishes with the organ, excess organ will be given to the research team for experimentation. In cases of recipient organs being removed for transplantation, they will be preserved in a plastic bag and then placed in the refrigerator. All experimentation will take place in the CRCHUM TID lab or Room 13 of the CHUM operating room.

Device insertion will occur with the designated needles and through the appropriate organ-specific route and imaging guidance. Multiple STING-MARK fiducials will be inserted. Plain film x-rays in 3 planes of the organs with the marker inserted will be taken and recorded.

Following experimentation, the organs will be appropriately labelled and returned to the pathology laboratory at the CHUM.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical resection of solid organs
* Recipients of solid organ transplantation

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Gain experience with deployability of the device in multiple organs, through different needles and different routes of insertion (trans-cutaneous, endoscopic). | Through study completion, an average of 1 year
  1) The deployability of the device will be measured with a deployability performance score (3=best over all metrics, 9=worst over all metrics) and compared with that of competing devices (Ultra EchoTip, Lumicoil) tested in parallel by the same user(s). No health outcomes are used in this score. Metrics used to establish this score are : operational efficiency ratio (the number of occurences of proper travel/anchoring/detaching over the total number of trials), time of operation and number of steps (from the first handling of the device to its detachment or lack thereof). Tests will be conducted on different organ locations (lung, oseophagus) with different routes of insertion (trans-cutaneous, endoscopic) using different models of 22Ga biopsy needles.
Verify stability of the device once inserted. | Through study completion, an average of 1 year
  2) The stability of the device after insertion will be measured with a stability performance score (3=best over all metrics, 9=worst over all metrics) and compared with that of competing devices (Ultra EchoTip, Lumicoil) tested in parallel by the same user(s). No health outcomes are used in this score. Metrics used to establish this score are mean three-dimensional fiducial displacement and maximal unidirectional displacement (along with its axis). These metrics are calculated by constructing a displacement vector map based on X-ray images of marker position relative to each other and to key neighbouring biological structures (tumor, bones, organs, other markers) taken each day over a period of 3 days.
verify radio-opacity of the device following insertion. | Through study completion, an average of 1 year
  3) The radio-opacity of the device after insertion will be measured with a stability performance score (4=best over all metrics, 12=worst over all metrics) and compared with that of competing devices (Ultra EchoTip, Lumicoil) tested in parallel by the same user(s). No health outcomes are used in this score. Metrics used to establish this score are : visual identification by surgeons and radiologists (based on their expertise by a simple yes/no criterion), automated radiotherapy machine software detection (based on the built-in detection criterion), mean pixel intensity and signal-to-noise ratio (from computer-based image analysis). These metrics are measured on MRI/X-ray/CT-scan images taken right after insertion and 1 day after insertion.

SECONDARY OUTCOMES:
User feedback regarding usability of the device | Through study completion, an average of 1 year
  Throughout all previsouly measured ouctomes, users will be asked to fill standard usability questionnaire SUS (10 questions, 0-100 score, >68 being considered above average). At the end of the experiments, users will be asked to fill a post-study usability questionnaire PSSUQ (16 questions, 1-7 score for each question, the lower the score, the better the performance and satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, Principal Investigator — CHUM
Locations (1):
- CHUM, Montreal, Quebec, Canada